CLINICAL TRIAL: NCT07144228
Title: Validation of a Platelet Proteomic Assay for Diagnosing and Monitoring Prostate Cancer: A Prospective Study.
Brief Title: Validation of a Platelet Proteomic Assay for Diagnosing and Monitoring Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Hessian Labs Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00116819
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer (Diagnosis)
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Control Group: Researchers are screening men who are suspicious of Pca, so those who will be negative for cancer will be the control group.
  Interventions: Device: HeLP TM
- Case Group: Researchers are screening men who are suspicious of Pca, so those who will be diagnosed will be the case group.
  Interventions: Device: HeLP TM

INTERVENTIONS:
Device: HeLP TM — lab test for prostate cancer

SUMMARY:
This is a single center study evaluating whether a new blood test based on platelet proteins rather than plasma proteins can improve detection of prostate cancer and evaluate the degree of serious disease. Currently, doctors rely on multiple tests such as PSA, MRI scans and biopsies to do the same evaluation. Researchers are trying to see if HeLP™ can be a safe and accurate alternative.

The study is inviting men who are being seen for suspicion of prostate cancer (based on symptoms or previous lab results). If they agree to be in the study, the research team will take a sample of their blood at the time they are getting a repeat PSA test or having Imaging. The research test does not affect the care they are already receiving and takes 3 extra tubes of blood (~3 tbsp).

The research team is aiming to include 300 participants total. They believe 278 people are needed to confidently compare results between people with and without prostate cancer.

They will do an interim analysis halfway through the study, once samples from 150 subjects have been collected.

The research is considered low risk-no more uncomfortable or dangerous than a blood draw. There is a risk of loss of privacy, but researchers are taking strong steps to protect privileged information. That includes proper data handling, secure, storage, and making sure the study team is trained in research ethics.

ELIGIBILITY:
Eligibility criteria

* Patients ≥ 40 years of age
* All patients with suspicion of PCa

Men ≥ 40 years of age attending Duke Health/Urology with suspicion of prostate cancer (Primary disease) will be approached to consent for the study. Upon consent, samples will be obtained alone, during repeat PSA/other biomarkers testing, or during imaging at Duke Lab.

Exclusion criteria

* Men who have previously undergone treatment for prostate cancer.
* Men with prior diagnosis of prostate cancer.
* Men with severe, irreversible coagulopathy.
* Men on anticoagulant therapies or those who have taken antiplatelet agents such as aspirin, NSAIDs (ibuprofen, entrophen, naproxen, diclofenac etc), clopidrogel, prasugrel, ticagrelor, or dipyridamole in the 7 days preceding blood collection.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is not relevant to women.
Study Population: All subjects meeting eligibility criteria will be offered participation in this research study. The study is not relevant to women. The terminally ill subjects, students, children or volunteers-will not be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Levels of HeLP™ proteins in the platelets of patients suspected to have PCa | Baseline
  Researchers will define the levels of HeLP™ proteins in the platelets of patients suspected to have PCa based on assessment within Duke Health compared to standard of care like PSA, mpMRI PI-RADS and other biomarkers (if available).
Diagnostic accuracy as reported by area under the curve (AUC) | Baseline
  Overall diagnostic accuracy of clinical variables including PSA, PI-RADS scoring, Hessian Map and other biomarkers (if available) will be determined and compared using receiving operating curve/area under curve analysis.

IPD SHARING:
Plan to Share IPD: No